CLINICAL TRIAL: NCT04447924
Title: The Effect of Daily Intake of Bifidobacterium Breve Bif195 on Small-intestinal Damage Induced by Ibuprofen - a Randomized, Double-blind, Placebo-controlled Trial in Healthy Volunteers.
Brief Title: The Effect of a Probiotic Strain on Ibuprofen-induced GI Damage
Acronym: PIP-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-GI-038
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Reduction of Small Intestinal Ulceration Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): Placebo arm. Similar trial product, but without Bif195 bacteria
  Interventions: Other: Placebo
- Bif195 arm (Experimental): Active trial product with minimum 15 billion CFU daily dose
  Interventions: Dietary Supplement: Bif195

INTERVENTIONS:
Dietary Supplement: Bif195 — Daily intake of Bif195 dietary supplement
  Arms: Bif195 arm
Other: Placebo — Daily intake of Placebo
  Arms: Placebo arm

SUMMARY:
To investigate if a daily dose of minimum 15 billion CFU of Bif195 reduces the risk of small-intestinal tissue damage in an Ibuprofen challenge model as assessed by video capsule endoscopy in a healthy US population.

DETAILED DESCRIPTION:
This trial is a single-site, randomized, double-blind, placebo-controlled, two-armed, parallel-group trial in healthy volunteers aged 18 - 40 years. The trial will investigate the effect of daily intake of the probiotic strain Bif195 or placebo when co-administered to daily intake of 800mg of Ibuprofen.

The trial includes a run-in period of two weeks duration followed by a six weeks intervention period where Bif195/placebo and Ibuprofen is co-administered.

Subjects will participate in the trial for a total duration of 8 weeks including the run-in phase. Besides the screening visit, the trial will consist of 5 visits.

After having given their written informed consent, subjects will complete the screening procedures to evaluate their eligibility for participation in the trial and complete a run-in period of two weeks duration to washout possible pre-trial probiotics and/or use of medication. After baseline assessments at Visit 2, subjects will start daily intake of 800mg of Ibuprofen and also be randomly assigned to 6-weeks daily intake of Bif195 or placebo product in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy and without any gastrointestinal pain or other significant symptoms
* Age 18 - 40 years
* Willing to abstain from any other probiotic products and/or medication known to alter gastrointestinal function throughout the participation of the trial

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Lewis score area-under-the-curve for Bif195 vs Placebo | 6 weeks
  The effect of Bif195 versus placebo on small intestinal mucosal damage during a 6-week Ibuprofen challenge measured as the area-under-the-curve of the Lewis scores obtained from all video capsule endoscopies between Visit 2 (randomization) and Visit 6 (end of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Eamonn Quigley, Professor, Principal Investigator — Houston Methodist Gastroenterology Associates
Locations (1):
- Atlantia Food Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No